CLINICAL TRIAL: NCT00330187
Title: Combined Pharmaco/Behavior Therapy in Adolescent Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kevin Gray, MD, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA17460; R01DA017460 (NIH)
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Nicotine Dependence; Nicotine Use Disorder
Keywords: nicotine dependence; bupropion SR; smoking cessation; adolescents; contingency management
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Bupropion SR + Contingency Management (Experimental): Bupropion SR capsules, with goal dose of 300 mg/day, for 6 weeks of treatment. Contingency Management, with escalating rewards for abstinence (and re-sets for non-abstinence) at twice-weekly visits.
  Interventions: Drug: Bupropion SR; Behavioral: Contingency Management
- Placebo + Contingency Management (Active Comparator): Placebo capsules, matched in appearance to Bupropion SR capsules, for 6 weeks of treatment. Contingency Management, with escalating rewards for abstinence (and re-sets for non-abstinence) at twice-weekly visits.
  Interventions: Behavioral: Contingency Management; Other: Placebo
- Bupropion SR + No Contingency Management (Active Comparator): Bupropion SR capsules, with goal dose of 300 mg/day, for 6 weeks of treatment. Contingency Management is not provided in this arm.
  Interventions: Drug: Bupropion SR
- Placebo + No Contingency Management (Placebo Comparator): Placebo capsules, matched in appearance to Bupropion SR capsules, for 6 weeks of treatment. Contingency Management is not provided in this arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupropion SR — Bupropion SR, with goal dose 300 mg/day, for 6 weeks of active treatment
  Arms: Bupropion SR + Contingency Management; Bupropion SR + No Contingency Management
Behavioral: Contingency Management — Contingency Management provided at twice-weekly visits during the 6-week active treatment. Escalating schedule, with resets, reinforcing smoking abstinence.
  Arms: Bupropion SR + Contingency Management; Placebo + Contingency Management
Other: Placebo — Placebo, matched in appearance to Bupropion SR, for 6 weeks of treatment
  Arms: Placebo + Contingency Management; Placebo + No Contingency Management

SUMMARY:
In the current proposal, we intend to study the efficacy of bupropion SR with or without combined contingency management (CM) among adolescent cigarette smokers. The proposed study will test not only medication (bupropion SR), but also combination of medication and CM in potentially improving smoking cessation outcomes AND retention of adolescent smokers in the study.

Hypothesis to be tested: Bupropion SR treatment will increase abstinence from cigarette smoking (as measured by urine cotinine and continuous abstinence) in adolescent smokers as compared to treatment with placebo only.

Hypothesis to be tested: Adolescent smokers treated with combined bupropion SR + contingency management (CM) treatment will have increased retention and increased abstinence rates when compared to bupropion SR alone or CM + placebo treated groups (as measured by decreased drop-out of participants, urine cotinine and continuous abstinence).

Hypothesis to be tested: CM will increase the abstinence from cigarette smoking (as measured by urine cotinine and continuous abstinence) in adolescent smokers as compared to treatment with placebo only.

DETAILED DESCRIPTION:
To test the hypotheses, 216 adolescent smokers will be recruited. Fifty-four adolescent smokers will be recruited in each of the four groups: bupropion SR only, bupropion SR + CM, CM + placebo, and placebo only. The cells will be balanced for gender and attention deficit hyperactivity disorder using permuted block randomization. A counseling intervention was added for all groups because it was reasoned that it would be unethical not to provide an active treatment to cigarette smoking adolescents. The counseling intervention will consist of two quit smoking brochures that provide information on tips to help quit smoking.

The study will consist of a one-week lead in period followed by a six-week treatment trial. For the medication groups, medications will be titrated during the one-week lead-in period. The primary outcome measure is urine cotinine and self-report of cigarette use collected using the Time-Line Follow-Back at the end of six weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Regular cigarette smokers smoking at least 5 cigarettes per day as derived by Time-Line Follow-Back method (Sobell et al., 1988). Average number of cigarettes per day (over past 30 days) will be used. Five cigarettes per day may seem low, but based on previous studies, adolescents tend to smoke fewer cigarettes per day as compared to adults.
2. Baseline urine cotinine level greater than 100 ng/ml.
3. Age range of 12 - 21
4. If under 18 yr. of age, parent(s) or guardian(s) able to participate in informed consent and initial assessment, or the participant must provide evidence of emancipated status.
5. For post menarchal female participants: agree to use birth control to avoid pregnancy.

Exclusion Criteria:

1. Active substance abuse/dependence (other than nicotine) within 2 weeks prior to participating in the study
2. Lifetime bipolar affective disorder (BPAD), psychosis, eating disorders. Bupropion may have adverse consequence on participants with these psychiatric diagnoses.
3. Current major depressive disorders. Since bupropion is also an antidepressant, this criteria is to minimize the confound of depressive disorder during the study. History of depressive disorders and current attention deficit hyperactivity disorder (ADHD) will not be an exclusion. We will use permuted block randomization procedure to balance the groups for ADHD.
4. Pregnancy or lactation. The safety of bupropion in pregnancy and during lactation is not well studied.
5. History of seizure disorder or predisposition to seizures (e.g., history of significant head trauma, currently taking medications that lower seizure threshold), since bupropion can lower seizure threshold.
6. History of severe renal, hepatic, neurological, or chronic pulmonary disease. This criterion was chosen due to the hepatic metabolism of bupropion.
7. Unstable medical problems
8. Allergy to bupropion
9. Current treatment with any other medication containing bupropion
10. Current treatment with any monoamine oxidase (MAO) inhibitors currently or within 2 weeks of starting the study since there may be serious and severe medical interactions between MAO inhibitors and bupropion SR.
11. Current treatment with nicotine replacement therapy (NRT)
12. History of intolerance or non-response to bupropion SR.
13. Current (past month) suicide ideation
14. Suicide attempt (past year)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himanshu P Upadhyaya, MS, MBBS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Gray KM, Carpenter MJ, Baker NL, Hartwell KJ, Lewis AL, Hiott DW, Deas D, Upadhyaya HP. Bupropion SR and contingency management for adolescent smoking cessation. J Subst Abuse Treat. 2011 Jan;40(1):77-86. doi: 10.1016/j.jsat.2010.08.010. Epub 2010 Oct 8. PMID 20934835

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupropion SR + Contingency Management | Placebo + Contingency Management | Bupropion SR + No Contingency Management | Placebo + No Contingency Management
Started | 37 | 36 | 29 | 32
Completed | 17 | 18 | 11 | 18
Not Completed | 20 | 18 | 18 | 14
Not completed — Lost to Follow-up | 12 | 13 | 14 | 10
Not completed — Withdrawal by Subject | 8 | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion SR + Contingency Management | Placebo + Contingency Management | Bupropion SR + No Contingency Management | Placebo + No Contingency Management | Total
Number analyzed (Participants) | 37 | 36 | 29 | 32 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 16 | 14 | 15 | 62
  Between 18 and 65 years | 20 | 20 | 15 | 17 | 72
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.4 (1.9) | 18.4 (1.9) | 18.1 (1.9) | 19 (1.8) | 18.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 11 | 15 | 56
  Male | 21 | 22 | 18 | 17 | 78

OUTCOME MEASURES:

1. Primary Outcome: Biologically-verified 7-day Point Prevalence Smoking Abstinence
Description: Self-reported abstinence for the past 7 days, confirmed by urine cotinine ≤100 ng/mL
Time Frame: End of treatment (week 6)
Population: Intent-to-treat analysis
Measure: Number; unit: participants
Arm/Group | Bupropion SR + Contingency Management | Placebo + Contingency Management | Bupropion SR + No Contingency Management | Placebo + No Contingency Management
Number analyzed (Participants) | 37 | 36 | 29 | 32
participants | 10 | 3 | 3 | 3
Statistical Analysis 1: Comparison: Bupropion SR + Contingency Management vs Placebo + No Contingency Management; Test type: Superiority; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 3.6, 95% CI 2-sided [0.9 to 14.4]

ADVERSE EVENTS:
Time Frame: Full study period (randomization through week 12 post-treatment follow-up visit)
Arm/Group | Bupropion SR + Contingency Management | Placebo + Contingency Management | Bupropion SR + No Contingency Management | Placebo + No Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/36 | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36 | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 22/37 | 14/36 | 25/29 | 15/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion SR + Contingency Management (N=37) | Placebo + Contingency Management (N=36) | Bupropion SR + No Contingency Management (N=29) | Placebo + No Contingency Management (N=32)
Headache (Nervous system disorders) | 12 (12) | 5 (5) | 6 (6) | 5 (5)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 9 (9) | 5 (5)
Irritability (Psychiatric disorders) | 8 (8) | 3 (3) | 5 (5) | 0 (0)
Vivid dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 8 (8) | 0 (0)
Other (General disorders) | 4 (4) | 6 (6) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes